CLINICAL TRIAL: NCT01515852
Title: General Anesthesia vs. Local Anesthesia in Stereotaxy
Acronym: GALAXY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Lutz Weise, Lutz Weise, M. D. Goethe University, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: JohannWGUH_GALAXY
Record Dates: First submitted 2012-01-23; First posted 2012-01-24 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Brain Lesion, Stereotactic Biopsy
Keywords: stress level; stereotactic biopsy; brain lesion; general anesthesia; local anesthesia
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress level after general anesthesia (Other)
  Interventions: Procedure: general anesthesia in stereotactic biopsy
- Stress level after local anesthesia (Other)
  Interventions: Procedure: local anesthesia in stereotactic biopsy

INTERVENTIONS:
Procedure: general anesthesia in stereotactic biopsy — stereotactic biopsy
  Arms: Stress level after general anesthesia
Procedure: local anesthesia in stereotactic biopsy — stereotactic biopsy
  Arms: Stress level after local anesthesia

SUMMARY:
Examination of stress level in general anesthesia in comparison to local anesthesia in stereotactic biopsy

DETAILED DESCRIPTION:
Stereotactic biopsy is routinely performed under local or general anesthesia. The advantage of local anesthesia might be reduction in cardiac and pulmonal complications, reduction of surgical time, and reduction of hospital stay. On the other hand it has been postulated that intraoperative seizures are avoided by general anesthesia and that brain tumor surgery is perceived in the public as psychological and physical stress.Therefor we postulate that patients undergoing stereotactic biopsies in local anesthesia show a higher stress level than patients operated under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* planned stereotactic biopsy
* age > 18 years

Exclusion Criteria:

* pregnancy
* anxiety disorder
* impaired consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
PTSS-10 | Three days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Johann Wolfgang Goethe University, Frankfurt am Main, Germany